CLINICAL TRIAL: NCT03648463
Title: Effect of Surgical Intervention on Mesenchymal Stem Cell Survival in Soft Tissue Reconstructive Procedures Using a Novel MRI Labeling Technique
Brief Title: Use of MRI Labeling Technique to Track Mesenchymal Stem Cell Survival in Orthopaedic Conditions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-46711
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Cartilage Degeneration; Rotator Cuff Tear; Osteoarthritis, Knee
MeSH Terms: conditions — Rotator Cuff Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not know if they received the surgical intervention that entails removing of the calcified cartilage or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthroscopy with removal of calcified cartilage (Experimental): This arm will have patients who will get surgical intervention (menisectomy, synovectomy and debridement) along with removal of the calcified cartilage layer. The patients will also get 5 cc of BMAC produced from The Harvest/Terumo BCT system.
  Interventions: Procedure: arthroscopy of the affected knee/ Bone Marrow Concentrate Injection
- arthroscopy without removal of calcified cartilage (Active Comparator): This arm will have patients who will get surgical intervention (menisectomy, synovectomy and debridement) but with retention of the calcified cartilage cap. The patients will also get 5 cc of BMAC produced from The Harvest/Terumo BCT system.
  Interventions: Procedure: arthroscopy of the affected knee/ Bone Marrow Concentrate Injection

INTERVENTIONS:
Procedure: arthroscopy of the affected knee/ Bone Marrow Concentrate Injection — Subjects will undergo knee arthroscopy for debridement, menisectomy and synovectomy of the cartilage defects. Subjects will also be injected with bone marrow aspirate concentrated harvested from the pelvis and centrifuged (produced produced using the Harvest/Terumo BCT system)
  Other Names: Injection of bone marrow aspirate concentrate harvested from the patient's iliac crest (produced using the Harvest/Terumo BCT system)

SUMMARY:
The primary objective is to determine whether a surgical intervention involving removing of the calcified cartilage cap in patients with Grade II Kellgren-Lawrence osteoarthritis influences the incorporation of labeled bone marrow aspirate concentrate (BMAC)-derived cells within the cartilage regenerate vs labeled BMAC cells delivered after arthroscopy without removing of the calcified cartilaginous layer. The survival and incorporation of the BMAC labeled cells will be evaluated with MRI using the Ferumoxytol infusion stem cell labeling technique. The second arm of the study evaluating cell fate after injecting stem cells under a rotator cuff repair will also be explored.

The secondary objectives are to 1) determine which surgical intervention leads to better clinical outcomes as measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) at 12 months, and 2) determine who long we can track the labeled-BMAC cells in the knee.

DETAILED DESCRIPTION:
Articular cartilage repair and regeneration has become a focal point for scientists and surgeons in search for a biological treatment for osteoarthritis that has failed non-operative management. Surgeons have begun to harvest and centrifuged bone marrow aspirate to produce bone marrow aspirate concentrate (BMAC) in hopes that the mesenchymal stem cells in the bone marrow aspirate can stimulate cartilage regeneration in areas of articular cartilage deficiency. This study is a first-in-human blinded randomized clinical trial using labeled BMAC cells in adults diagnosed with grade II-III Kellgren-Lawrence osteoarthritis.

This is a single site study where 20 cases among eligible patients will be identified and randomly assigned to either the control (no calcified cartilage) or experimental (calcified cartilage removed) group. A power analysis will be performed after 20 patients to determine the total number of patients required to reach adequate power.

A patient will receive an infusion of Feraheme 2 days before the procedure and a baseline MR Pelvis and knee. A nurse will be present at all times during the infusion to monitor vitals. On the day of the procedure patient will undergo harvesting of the bone marrow from the pelvis and arthroscopy procedure involving menisectomy, synovectomy and debridement. Patients in the experimental group will also undergo removal of the calcified cartilage cap. The bone marrow aspirate will be centrifuged and about 5-7 cc of BMAC injected into knee. MRIs will be done at the 2 day mark for confirmation of the labeling of the mesenchymal cells, and at the two week and 3 month mark. Patient related Outcomes will be measured using the Knee injury and Osteoarthritis Score at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 30-70 patients with Kellgren grade II-III osteoarthritis,
2. Symptomatic knee pain greater than 6 months
3. At least one discrete contained chondral defect
4. Failed a minimum of 6 weeks of physical therapy
5. Grossly normal knee alignment: <5 degrees of varus or valgus alignment
6. Lesion located on medial or lateral femoral condyle or trochlea

Exclusion Criteria:

1. Radiographs demonstrating either no or little osteoarthritis (Kellgren-Lawrence Grade 0 or 1)
2. Diagnosis of Inflammatory (RA, JIA etc) or infectious arthritis
3. Malalignment of mechanical axis > or = 5 degrees of varus/valgus
4. Cortisone and/or Hyaluronic acid intra-articular injection within the last 3 months
5. Ligamentous knee instability
6. The subject is on ongoing specific osteoarthritis drugs such as chondroitin sulphate, diacerein, N-glucosamine, piascledine, capsaicin in the 2 weeks prior to baseline treatment
7. BMI > 30
8. Currently pregnant or planning to become pregnant (no MRI possible).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Integration of the mesenchymal stem cells. | 3 months
  Number of integrated labeled mesenchymal stem cells in the cartilage regenerate counted from from MRI imaging.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (pain subscale) | 12 months
  KOOS pain score at baseline and at 12 months to measure functional outcomes. This sub scale of the KOOS questionnaire has a possible total of 100 points (higher scores mean less pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Enweze, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Undecided